CLINICAL TRIAL: NCT02951299
Title: Branch Director, Division of Nephrology, Department of Internal Medicine, Taipei Medical University Hospital.
Brief Title: The Protective Effect of Pentoxifylline on Acute Kidney Injury
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hsi-Hsien Chen, Medical attending, Taipei Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201507004; 104-TDU-B-212-113001 (Other Grant/Funding Number: MOHW)
Record Dates: First submitted 2016-10-25; First posted 2016-11-01 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-11

CONDITIONS: Pentoxifylline; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Pentoxifylline; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pentoxifylline group (Experimental): Received oral pentoxifylline (400 mg) three times a day for 14 days.
  Interventions: Drug: Pentoxifylline 400Mg Tablet
- no treatment group (No Intervention): No intervention.

INTERVENTIONS:
Drug: Pentoxifylline 400Mg Tablet — Investigators with AKI will received oral pentoxifylline (400 mg) three times a day for 14 days or no pentoxifylline according to their decision.
  Arms: pentoxifylline group

SUMMARY:
Acute kidney injury (AKI) has a frequency of 7.0 % in hospital inpatients and is especially common in critically ill patients, in whom the prevalence of acute kidney injury is greater than 40% at admission to the intensive care unit if sepsis is present. Therefore, alternative strategies are required to confer better or more complete renoprotection for those who suffered from AKI.

There had been many studies demonstrated that the phosphodiesterase inhibitor pentoxifylline (PTX) is a potent anti-inflammatory, anti-proliferative, and anti-fibrotic agent capable of attenuating experimental renal disease such as drugs, ischemic and sepsis induced AKI. We thereby design this controlled, non-randomized clinical trial, aiming at investigating the potential renoprotective efficacy of PTX, as compared to placebo, in 200 patients with AKI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) refers to a clinical syndrome characterized by a rapid (hours to days) decrease in renal function, which is a common and important diagnostic and therapeutic challenge for clinicians. The disorder has a frequency of 7.0 % in hospital inpatients and is especially common in critically ill patients, in whom the prevalence of acute kidney injury is greater than 40% at admission to the intensive care unit if sepsis is present. AKI is independently associated with important morbidity and mortality although many efforts have been used in past years. Therefore, alternative strategies are required to confer better or more complete renoprotection for those who suffered from AKI.

There had been many studies demonstrated that the phosphodiesterase inhibitor pentoxifylline (PTX) is a potent anti-inflammatory, anti-proliferative, and anti-fibrotic agent capable of attenuating experimental renal disease such as drugs, ischemic and sepsis induced AKI. We thus hypothesized that PTX may have therapeutic value for AKI in human. We thereby design this controlled, non-randomized clinical trial, aiming at investigating the potential renoprotective efficacy of PTX, as compared to placebo, in 200 patients with AKI.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 ~ 70 y/o who had admitted for acute kidney injury (renal function decreased within 48hours which meets following criteris: GFR decreased > 25 %, serum creatinine elevated > 0.3 mg/dl or 50%、urine amount less than 0.5 ml/kg/hour > 6 hours).

Exclusion Criteria:

* 1. Those who had been received regular dialysis or GFR < 30 ml/min before test. 2. Those who with acute bleeding. 3. Those who allergy to pentoxifylline or methylxanthine derivatives (such as caffeine, theophylline and theobromine )..

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2017-06-01 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Renal outcome | 4 weeks
  Need of dialysis

SECONDARY OUTCOMES:
Renal function tests | 4 weeks
  Serum and urine test (Blood urine nitrogen, Serum creatinine, Daily urine amount)
inflammation marker | 4 weeks
  Transforming Growth Factor-β; Monocyte chemoattractant protein-1

IPD SHARING:
Plan to Share IPD: No